CLINICAL TRIAL: NCT02730273
Title: The Evaluation of a Nasal Mask for the Treatment of Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-184
Record Dates: First submitted 2016-03-13; First posted 2016-04-06 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial Nasal Mask (Experimental): Participants to use nasal mask in-home for a week and one night in lab overnight polysomnography.
  Interventions: Device: Trial Nasal mask

INTERVENTIONS:
Device: Trial Nasal mask — Nasal mask for the treatment of obstructive sleep apnea (OSA)

SUMMARY:
This investigation is designed to evaluate the performance (leak and comfort) as well as the participant's overall acceptance of the trial nasal mask amongst Obstructive Sleep Apnea (OSA) participants. An important factor in this investigation will be the testing of two different seal sizes on the participants (medium and large size). A total number of 12 participants who currently use nasal or nasal pillow masks will be recruited for the trial. Participants have been selected based on their anthropometric measurements collected in previous trials (CIA-103). Participants from previous NZ trials may be recruited into this trial with their consent. All the participants will be recruited from the Fisher & Paykel Healthcare Database of subjects with OSA (Ethics Reference NTY/08/06/064), Auckland District Health Board (ADHB) and New Zealand Respiratory and Sleep Institute (NZRSI).

Participants will use the trial mask in home for a period of 7 ± 3 days and also 1 overnight polysomnography session at the Fisher & Paykel Healthcare sleep lab. Baseline data will be collected from the participant during the first visit, 7 days of CPAP usage data will be downloaded and stored for analysis. The participant will use the trial device on their usual Continuous or Auto Positive Airway Pressure (CPAP/APAP) setting and device for the duration of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Able to give consent
* Apnea Hypopnea Index (AHI) ≥ 5 on diagnostic night
* Prescribed a Continuous Positive Airway Pressure (CPAP) device after successful OSA diagnosis
* Existing nasal or nasal pillow mask user

Exclusion Criteria:

* Inability to give consent
* Patients who are in a coma or a decreased level of consciousness.
* Anatomical or physiological conditions making APAP therapy inappropriate (e.g. unconsolidated facial structure)
* Commercial drivers who are investigated by New Zealand Transport Agency (NZTA)
* Current diagnosis of CO2 retention
* Pregnant or may think they are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Objective leak data (L/min) | Up to 1 week in-home
  Obtained from the participant's device
Subjective measurement of leak | Up to 1 week in-home
  Subjective Questionnaire
Comfort | Up to 1 week in-home
  Subjective Questionnaire
Stability | Up to 1 week in-home
  Subjective Questionnaire
Draft | Up to 1 week in-home
  Subjective Questionnaire
Noise | Up to 1 week in-home
  Subjective Questionnaire
Objective leak data (L/min) | 1 night
  Obtained from the overnight polysomnography

SECONDARY OUTCOMES:
Preference of the mask | Up to 1 week in-home
  Subjective Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kayan Gonda, BSc, Principal Investigator — Sponsor Employee
Locations (1):
- Fisher & Paykel Healthcare, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
For product development purposes only. Data will be deidentified.